CLINICAL TRIAL: NCT05735574
Title: To Determine the Cost of Explant and Management of Spinal Cord Stimulation Devices Related to Implantable Pulse Generator Infection in a Single Center Specializing in Neuromodulation
Brief Title: Determining Cost of Explant of Neurmodulation Device Due to Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 307575
Record Dates: First submitted 2023-01-26; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Neuropathic Pain; Infections; Device Related Sepsis; Chronic Pain
Keywords: Spinal Cord Stimulation; Neuromodulation
MeSH Terms: conditions — Neuralgia; Infections; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IPG infections — Infected IPGs
  Other Names: Infected IPG

SUMMARY:
Spinal cord stimulation (SCS) is a medical device inserted beside the spine to treat nerve pain. When the device becomes infected (which happens 4 % of the time) it needs to be taken out and put back in again at a later date. So far we are unsure of how much this process costs. I am going to analyse data collected on a database of all devices taken out due to infection and calculate an average cost of taking them out, the intermediate care and putting them back in again in our hospital only. This will enable us to understand how much this process costs and if there are any methods of reducing the chance of infection in the future; we will be able to work out how much the NHS should pay for these products based on this data. This will be done in Guys and St Thomas's from a database in the chronic pain research department in patients who had their device taken out due to infection. It will take 6 months and will all be retrospective. Additional details may be collected from patients electronic records where needed. These will be collected by a member of the direct care team and pseudonymised prior to adding to the research data set.

DETAILED DESCRIPTION:
Design: Retrospective chart and electronic record review of all explants due to infection with cost analysis up to re-implantation.

Methods:

Based on a database there are approximately N=18-20 infections over 7 years with adequate data to determine the overall cost of explant due to infection. The data to be collected will include: hospital admission, surgical time, blood tests, swabs, antibiotic therapy, additional outpatient visits, cost of re-implantation. These can be collected from electronic patient records (EPR). The cost of individual patient admissions will be obtained from the account services at Guys and St Thomas's and sent in a password protected database.

The site of infection will also be recorded and this can be obtained from the operative note. A study by Hayek and colleagues have indicated only 10% of infections are at the lead site and the majority are at the IPG site. Another review by Follet and colleagues have indicated only 54% of infections are at the IPG site, 17% at the lead site and the others not clearly determined. For this reason, there will need to be a range of costs based on the confirmed and the indeterminate sites of infection. The main focus of this paper will be on IPG infections since TYRX is only used at the IPG site.

Economic metrics will also be taken into consideration which have been described in the UK as some patients for technical reasons cannot be re-implanted with SCS systems after infection. The cost effectiveness of this therapy is essentially lost in these patients forever. The time proceeding to re-implantation can also be reviewed and incorporated. There was an NIHR review of cost analysis of these systems published in the UK that can be used for this. Specifically the cost of SCS and conventional medical management (CMM) is £3440 in year one of these devices and CMM alone is £6936.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who had an explant of a neuromodulation device due to infection between 2013-2020 in our centre.
* Any patient who had as suspected explant of a spinal cord stimulator due to infection

Exclusion Criteria:

• Explant of a device for another reason

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that have neuromodulation devices explanted due to infection
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Cost of explant, intermediate care and re-implantation of device | Until device re-implanted which will vary from 3 months- 1 year
  Cost of explant, intermediate care and re-implantation of device

SECONDARY OUTCOMES:
Pathway of patients from device explantation until re-implantation of device | up to re-implant or decision not to which will vary from 3 month- 1 year

IPD SHARING:
Plan to Share IPD: No
There will only be a report to the financial sponsor in anonymous format

REFERENCES:
- [Result] Al-Kaisy A, Royds J, Al-Kaisy O, Palmisani S, Pang D, Smith T, Padfield N, Harris S, Wesley S, Yearwood TL, Ward S. Explant rates of electrical neuromodulation devices in 1177 patients in a single center over an 11-year period. Reg Anesth Pain Med. 2020 Nov;45(11):883-890. doi: 10.1136/rapm-2020-101681. Epub 2020 Aug 26. PMID 32848088